CLINICAL TRIAL: NCT05709288
Title: A Pilot Study Evaluating the Safety, Tolerability and Efficacy of Gene Therapy With BBM-H901 in Hemophilia B Patients Aged 12-18 Years Old
Brief Title: Gene Therapy for Hemophilia B Patients Aged 12-18 Years Old
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022051
Record Dates: First submitted 2023-01-19; First posted 2023-02-02 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-01

CONDITIONS: Hemophilia B
Keywords: gene therapy; AAV
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Intervention Model Description: Hemophilia B patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BBM-H901 administration group (Experimental): Subjects will be administered with single dose intravenous infusion of BBM-H901.
  Interventions: Drug: BBM-H901

INTERVENTIONS:
Drug: BBM-H901 — Single dose intravenous infusion of BBM-H901, an adeno-associated viral (AAV) vector designed to drive expression of an hyper active human factor IX mutant(FIX Padua) transgene in liver. The dose of BBM-H901 is 5x10'12 vg/Kg.

SUMMARY:
This is a Phase 1, open- label, non- randomized, uncontrolled, single dose pilot study to evaluate the safety, tolerability and efficacy of a single intravenous infusion of BBM-H901 in hemophilia B subjects with ≤2IU/dl residual FIX levels and aged 12-18 years old. BBM-H901 is an adeno-associated viral (AAV) vector designed to drive expression of the human factor IX (hFIX) transgene and raise circulating levels of endogenous FIX.

DETAILED DESCRIPTION:
This is a Phase 1, open- label, non- randomized, uncontrolled, single dose pilot study to evaluate the safety, tolerability and efficacy of a single intravenous infusion of BBM-H901 in hemophilia B subjects with ≤2IU/dl residual FIX levels and aged 12-18 years old. BBM-H901 is an adeno-associated viral (AAV) vector designed to drive expression of the human factor IX (hFIX) transgene and raise circulating levels of endogenous FIX. Nine subjects will be enrolled and administered with single infusion of BBM-H901, an AAV at one dose level of 5x10'12 vg/Kg. Subjects and statutory guardian must provide informed consent and then undergo screening assessments up to 4-8weeks prior administration of BBM-H901. All subjects will undergo 52(+- 2) weeks safety observation and will be continuously followed up to evaluate long- term safety and efficacy of BBM-H901 up to ten years. The first subject will be dosed at 5x10'12 vg/Kg and undergo 8 weeks safety observation of which the data will undergo review by an independent safety committee.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects and statutory guardian must be able to understand the purpose and risks of the study and provide signed and dated informed consent;
2. Be male and 12≤ age <18 years of age, body wight ≥ 50kg;
3. Have hemophilia B with ≤2 IU/dL (≤2 %) endogenous FIX activity levels as documented by a certified clinical laboratory at the time of screening. If the screening result is >2% due to insufficient washout from FIX protein product, then the severity of hemophilia B may be confirmed by documented historical evidence from a certified clinical laboratory demonstrating ≤2% FIX coagulant activity (FIX:C) ;
4. Had had ≥75 prior exposure days (EDs) to any recombinant and/or plasma-derived FIX protein products based on historical data from the subject's record/history;
5. With ≤ 1:4 neutralizing antibodies and ≤1:200 binding antibodies against BBM-H901 capsid;
6. Subjects with bleeding episode and/ or FIX agents infusion events within 12 weeks prior to screening;
7. Have no prior history of hypersensitivity or anaphylaxis associated with any FIX or IV immunoglobulin administration;
8. Have no measurable FIX inhibitor as assessed by laboratory; or documented no prior history of FIX inhibitor (family history of inhibitors will not exclude the subject) and no clinical signs or symptoms of decreased response to FIX administration;
9. Have acceptable laboratory values:

   1. Hemoglobin ≥11 g/dL ;
   2. Platelets ≥100,000 cells/μL;
   3. AST, ALT ≤1.5x upper limit of normal at the testing laboratory;
   4. Bilirubin ≤1.5x ULN ;
   5. glomerular filtration rate eGFR ≥ 60ml/min.
10. For those subjects with sexual maturity, subject and statutory guardian must know that subjects must agree to use reliable barrier contraception until 52 weeks;
11. with good compliance to the schedule of visit and fill in the subject diary.

Exclusion Criteria:

1. Hepatitis B surface antigen antibody (HBSAg-Ab) or HBV-DNA positive; hepatitis C antibody or HCV-RNA positive;
2. Currently on antiviral therapy for hepatitis B or C;
3. With coagulation disorders other than hemophilia B;
4. Had immunosuppressive therapy other than steroid and other suggested IST agents within 30 days prior to screening;
5. Had vaccine 30 days prior to screening or have scheduled vaccination plan during the study (up to 52 weeks);
6. Have significant underlying liver disease, as defined by a preexisting diagnosis of portal hypertension, splenomegaly, encephalopathy, etc; other liver conditions unsuitable to gene therapy judged by investigator;
7. Have surgery plan within 52 weeks after gene therapy;
8. Have history of chronic infection or high rish of infection that the Investigator considers to constitute an unacceptable risk;
9. Had participated in a previous gene therapy research trial within the last 52 weeks or in a clinical study with an investigational drug within the last 12 weeks;
10. Had any herb that may affect the liver function within 4 weeks prior to screening;
11. Have history of fatal bleeding episode, eg intracranial hemorrhage, etc;
12. Any concurrent clinically significant major disease or any other condition that, in the opinion of the Investigator, makes the subject unsuitable for participation in the study;

Ages: 12 Years to 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2035-06 (Estimated); Study Completion 2035-11 (Estimated)

PRIMARY OUTCOMES:
The incidence of treatment related adverse events deemed related to BBM-H901 within 10 weeks after vector administration | infusion to 10 weeks after vector infusion.
  the type and incidence of TRAE after BBM-H901 infusion according to the CTCAE(v5.0)
The incidence of adverse events and serious adverse events within 52 weeks after BBM-H901 administration | Vector infusion to 52 weeks after gene therapy.
  Number of patients experiencing treatment-related adverse events from vector infusion to 52 weeks after vector infusion.
Change from baseline aspartate amino transferase | At multiple timepoints from pre-dose through up to 1 years post-dose
  number of subjects with elevation of AST. Number of episodes of elevating AST
Change from baseline alanine aminotransferase | At multiple timepoints from pre-dose through up to 1 years post-dose
  number of subjects with elevation of ALT. Number of episodes of elevating ALT

SECONDARY OUTCOMES:
Vector shedding after BBM-H901 infusion | multiple timepoints until 2 consecutive negative results achieved usually within 52 weeks
  Vector genome in plasma, urea, stool, saliva will be monitored
Vector derived Factor IX(FIX) activity | infusion to 52 weeks after gene therapy
  FIX:C measured using one- stage APTT based method
Annualized bleeding rate(ABR) after gene therapy | vector infusion to 52 weeks after gene therapy
  ABR will be prospectively collected at each visit.
Times of infusion of factor IX agents | vector infusion to 52 weeks after gene therapy
  Times of infusion of factor IX agents, eg FIX concentrates, prothrombin complex concentrate, fresh- frozen plasma.
number of target joint | vector infusion to 52 weeks after gene therapy
  target joint is defined as a joint with ≥bleeding during the last 6 months
factor IX inhibitor | vector infusion to 52 weeks after gene therapy
  factor IX inhibitor will be measured using bethesda method

OTHER OUTCOMES:
Long term factor IX activity | 52 weeks after gene therapy to up to 10 years
  factor IX activity will be measured using one stage APTT based method
Long term Annualized bleeding rate | 52 weeks after gene therapy to up to 10 years
  Annualized bleeding rate will be calculated based on the bleeding times and time interval

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Insitute of haematology and blood diseases hospital, chinese academy of medical sciences
Locations (1):
- Institute of haematology and Blood diseases hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Researchers qualified can request the dataset, including de-identified individual subject data. Data may be requested from PI from 12 months 36 months after study completion.
Supporting Information: Study Protocol
Time Frame: From 12 months 36 months after study completion.
Access Criteria: Upon request to PI.